CLINICAL TRIAL: NCT01962597
Title: Comparison of Aerobic Exercise, Strength Training, or Its Combination in Hemodialysis Patients: a Randomized Controlled Trial
Brief Title: Trial of Hemodialysis Based Exercise for Strength Improvement Study
Acronym: THESIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Scott Brimble, Staff Nephrologist/Associate Professor of Medicine, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-468
Record Dates: First submitted 2013-10-08; First posted 2013-10-14 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: End Stage Renal Disease
Keywords: hemodialysis; aerobic exercise; resistance training; walking speed; randomized controlled trial
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Exercise; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- aerobic exercise (Active Comparator): patients will undergo supervised exercise on a bike ergometer for 30 minutes three times per week during hemodialysis
  Interventions: Other: aerobic exercise
- resistance training (Active Comparator): patients will undergo supervised lower extremity strength training three times per week pre-hemodialysis
  Interventions: Other: resistance training
- aerobic exercise and resistance training (Experimental): patients will undergo a combination of aerobic exercise and resistance training on an alternating schedule three time per week
  Interventions: Other: aerobic exercise; Other: resistance training

INTERVENTIONS:
Other: aerobic exercise
  Arms: aerobic exercise; aerobic exercise and resistance training
Other: resistance training
  Arms: aerobic exercise and resistance training; resistance training

SUMMARY:
Study Hypothesis: The combination of aerobic and resistance exercise training will improve walking speed compared to either individual intervention.

Brief Summary:

Sixty hemodialysis participants who meet inclusion and exclusion criteria will be randomized to 20 weeks of supervised exercise, using either: (i) on-dialysis aerobic exercise using a bike ergometer; (ii) pre-dialysis leg strength training using weights; or (iii) both. The primary outcome is walking speed over 4-metres. Secondary outcomes will include:

(i) short physical performance battery; (ii) health-related quality of life [EuroQOL-5D-5L]; (iii) Dialysis recovery time; (iv) Nottingham extended activities of daily living (EADL) index; (v) Leg strength; (vi) body composition and anthropometry.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* On hemodialysis minimum of 3 times per week
* On hemodialysis > 3 consecutive months

Exclusion Criteria:

* Inability to provide consent
* Inability to walk 4-metres
* Chest pain with exertion or myocardial infarction in past 6-months
* Pre-dialysis systolic blood pressure > 200 mm Hg or diastolic BP > 100 mm Hg in past 2-weeks
* Functional or cardiorespiratory limitations preventing use of cycle ergometer for at least five-minutes or the ability to perform single maximum rep with each of resistance exercises described
* Joint replacement or lower extremity fracture in previous 6-months
* Severe cognitive impairment
* Currently using corticosteroids >5 mg/day
* Pre-dialysis serum potassium in previous month less than 3.5 or greater than 6.0 mmol/L.
* Attending nephrologist feels exercise is medically contraindicated
* Scheduled living related kidney transplant in next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-06 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
change in walking speed over 20 weeks | 10 and 20 weeks
  repeated measures analysis

SECONDARY OUTCOMES:
change in short physical performance battery over 20 weeks | 10 and 20 weeks
  repeated measures analysis
change in EuroQOL-5D-5L over 20 weeks | 10 and 20 weeks
  Health-related quality of life. Repeated measures analysis
change in dialysis recovery time over 20 weeks | 10 and 20 weeks
  repeated measures analysis
change in Nottingham extended activities of daily living index over 20 weeks | 10 and 20 weeks
  repeated measures analysis
change in body anthropometry and composition over 20 weeks. | 10 and 20 weeks
  weight, waist-hip ratio, bioimpedance analysis-determined fat-free mass, percentage body fat, phase angle. Repeated measures analysis
change in inflammation measures over 20 weeks | 10 and 20 weeks
  serum albumin, C-reactive protein, interleukin-6 and tumor necrosis factor-alpha. Repeated measures analysis
hospitalization | continuous over 20 weeks
death | continuous over 20 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- St. Josephs Healthcare Hamilton, Hamilton, Ontario, Canada